CLINICAL TRIAL: NCT03540914
Title: Effect of Acetazolamide on Right Heart Function at Rest in Lowlanders Older Than 40 Years at Altitude.: A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Right Heart Function at Rest in Lowlanders Older Than 40 Years at Altitude.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-01-8/305E
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Altitude Hypoxia
Keywords: healthy participants older than 40 years; right heart function; prevention; acetazolamide
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 1x125mg acetazolamide in the morning, 2x125mg in the evening, starting 24 hours before departure to 3'100m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3'100m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of acetazolamide on right heart function at rest in lowlanders older than 40 years travelling from 760 m to 3'100 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of preventive acetazolamide intake on right heart function at rest in lowlanders older than 40 years travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3'100 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo), will be administered before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3'100 m.

An interim analysis will be carried out when 200 participants will have completed the study and/or after the first year. The Peto's method will be used and the trial will be stopped when pre-specified futility boundaries were crossed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, age 40-75 yrs, without any disease and need of medication.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.
* Kyrgyz ethnicity

Exclusion Criteria:

* Any active respiratory, cardiovascular or other disease requiring regular treatment or being otherwise relevant for tolerance of hypoxia or altitude exposure.
* Any condition that may interfere with protocol compliance including current heavy smoking (>20 cigarettes per day or >20 pack-years with active smoking during the last 10 years), regular use of alcohol.
* Allergy to acetazolamide and other sulfonamides.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change of pulmonary artery pressure evaluated by echocardiography from 760 m baseline measurement to measurement at 3100 m in the acetazolamide compared to the placebo group | Day 2 at 760m and 3100m
  Difference in change of pulmonary artery pressure evaluated by echocardiography from 760 m baseline measurement to measurement at 3100 m between acetazolamide and placebo groups

SECONDARY OUTCOMES:
Difference in pulmonary artery pressure evaluated by echocardiography at 3100 m in the acetazolamide compared to the placebo group | Day 2 at 3100m
  Difference in pulmonary artery pressure evaluated by echocardiography at 3100 m in the acetazolamide compared to the placebo group
cardiac output | Day 2 at 760m and 3100m
  Difference in altitude-induced change of cardiac output between acetazolamide and placebo group, measured by transthoracic echocardiography
cardiac output | Day 2 at 3100m
  Difference at altitude between acetazolamide and placebo group in cardiac output, measured by transthoracic echocardiography
right heart dimensions | Day 2 at 760m and 3100m
  Difference in altitude-induced change of right heart dimensions between acetazolamide and placebo group, measured by transthoracic echocardiography
right heart dimensions | Day 2 at 3100m
  Difference at altitude of right heart dimensions between acetazolamide and placebo group, measured by transthoracic echocardiography
right heart function | Day 2 at 760m and 3100m
  Difference in altitude-induced change of right heart function between acetazolamide and placebo group, measured by transthoracic echocardiography (TAPSE)
right heart function | Day 2 at 3100m
  Difference at altitude of right heart function between acetazolamide and placebo group, measured by transthoracic echocardiography (TAPSE)
stroke volume | Day 2 at 760m and 3100m
  Difference in altitude-induced change of stroke volume between acetazolamide and placebo group, measured by transthoracic echocardiography
stroke volume | Day 2 at 3100m
  Difference at altitude between acetazolamide and placebo group in stroke volume, measured by transthoracic echocardiography
volumes | Day 2 at 760m and 3100m
  Difference in altitude-induced change of volumes between acetazolamide and placebo group, measured by transthoracic echocardiography
volumes | Day 2 at 3100m
  Difference at altitude of volumes between acetazolamide and placebo group, measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev,, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, MSc, Principal Investigator — University Hospital, Zürich; Silvia Ulrich, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Mayer L, Lichtblau M, Furian M, Buergin A, Saxer S, Mademilov M, Bader PR, Schneider SR, Sooronbaev T, Bloch KE, Ulrich S. Effect of Acetazolamide on Pulmonary Hemodynamics and Right Heart Function in Healthy Adults Going to Altitude: A Randomized Controlled Trial. J Am Heart Assoc. 2025 Sep 2;14(17):e041941. doi: 10.1161/JAHA.125.041941. Epub 2025 Aug 29. PMID 40878988